CLINICAL TRIAL: NCT00852774
Title: Effects of Steep Trendelenburg Positioning on Intra-Ocular Pressure During Surgery For Endometrial Cancer: Robotics Versus Laparotomy
Brief Title: Steep Trendelenburg Positioning on Intra-Ocular Pressure During Surgery for Endometrial Robotics Versus Laparotomy
Status: Withdrawn | Type: Observational
Why Stopped: terminated due to low staffing
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, David Cohn, Principal Investigator, Ohio State University
Other Study IDs: OSU-08159; NCT01375192 (obsolete NCT alias)
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Endometrial Cancer Patients Hysterectomy Robotic Surgery
- 2: Endometrial Cancer Patient Hysterectomy Laparotomy Surgery

SUMMARY:
The purpose of this study is to assess changes of intra-ocular pressure (IOP) and examine preoperative facts affecting IOP in endometrial cancer patients undergoing robotic hysterectomy compared to laparotomy.

DETAILED DESCRIPTION:
All patients that are surgical candidates with endometrial cancer will be screened for this study. Two measurements from each eye will be taken in the following positions: awake at rest, supine before induction, after induction on anesthesia, after insufflation of abdomen with CO2 in supine position, in trendelenburg position, in deep trendelenburg position,at the end of procedure,prior to awakening in supine position and one last reading 45-60 min after awakening in supine position. The time, blood pressure, heart rate, peak airway pressure, plateau airway pressure, end tidal desflurane, end tidal CO2, total IV fluids administered, and blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial Cancer Surgery

Exclusion Criteria:

* Not a surgical candidate

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endometrial Cancer Surgical Candidates
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To assess the changes in intra-ocular pressure and examine perioperative factors affecting IOP in endometrial cancer patients undergoing robotic hysterectomy compared to a laparotomy | 5years for enrollment completion

CONTACTS AND LOCATIONS:
Overall Officials: David Cohn, MD, Principal Investigator — Ohio State University